CLINICAL TRIAL: NCT04093063
Title: An Inexpensive Practice Model for Microsurgical Skills Training: A Randomized Trial
Brief Title: Validating an Inexpensive Practice Model for Microsurgical Skills Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Sangita Patel, Principal Investigator, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00001491
Record Dates: First submitted 2019-09-16; First posted 2019-09-17 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Microsurgery
Keywords: microsurgery; ophthalmology; medical education; surgical skills; surgical practice

STUDY DESIGN:
Intervention Model Description: This study is a single-center, prospective, randomized, controlled trial. After obtaining consent, recruited participants were asked to perform a microsurgical task. Their attempt was video-recorded for a pre-assessment. After completion of the video-recorded pre-assessment, participants were randomized to either the intervention or the non-intervention control group by flip of a coin. Subjects in the intervention group were tasked to build a micro-stellated icosahedron using a detailed instruction manual. Subjects in the control group had no specific task for two weeks.
  All subjects in both groups were required to return in two weeks for a second in-person meeting. At the second meeting, their attempt at completing a microsurgical task was video-recorded for a post-assessment, using similar instruments and set-up as those used two weeks prior.
Who Masked: Investigator, Outcomes Assessor
Masking Description: In order to judge the effectiveness of intervention, participants in the intervention and control groups will perform a microsuturing task at the beginning and at the end of the study to grade surgical skills. Before each grading session, subjects will watch video instructions on how to perform microsurgical suturing. The subjects' microsurgical manipulations will be video-recorded. The video-recordings will be rated by 2 ophthalmologists, including the main investigator, masked to the identity of the subject (intervention vs control) and time of recording (either before or after intervention). Videos were muted, and subjects were instructed to wear gloves in order to ensure anonymity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Subjects in the intervention group were tasked with building a micro-stellated icosahedron using a detailed instruction manual. They were each provided with a dissecting microscope and necessary materials to complete the task at home at their leisure. They were given two weeks to complete the task. They were asked to return for a second in-person meeting two weeks.
  Interventions: Other: Micro-stellated Icosahedron
- Control Group (No Intervention): Subjects in the non-intervention control group were not given any task or any materials. They were asked to return for a second in-person meeting in two weeks.

INTERVENTIONS:
Other: Micro-stellated Icosahedron — A portable, inexpensive microsurgery training model that requires the following materials for completion. a stereoscopic dissecting microscope, two jeweler style forceps, a pair of curved-tip micro scissors , 1 meter of monofilament nylon thread, 0.5 meter of polyimide microtubule material , one 15 cm metal ruler, a scalpel blade (#15), and double-sided tape. For a microsurgically-naive subject, a total of 20 hours are required to complete this model.
  Arms: Intervention Group

SUMMARY:
A single-center, prospective, randomized, controlled intervention trial to validate an inexpensive practice model for acquisition of microsurgical skills. Following a pre-assessment microsurgical skills task, participants were randomized to either an intervention group to build a micro-stellated icosahedron, or to a control group with no specific task assigned. A post-assessment microsurgical skills task was given to all participants after two weeks. Videos of pre- and post-assessments were masked and independently rated by two ophthalmologists using Video-based Modified Objective Structure Assessment of Technical Skill (OSATS) scoring criteria. Analyses were done to determine improvement in time required to complete tasks and in scores between pre- and post- assessments.

DETAILED DESCRIPTION:
This study is a single-center, prospective, randomized trial approved by the University at Buffalo Institutional Review Board. Medical students, residents and other interested individuals without prior microsurgery experience affiliated with the Jacobs School of Medicine and Biomedical Sciences were invited to participate. Each participant completed written informed consent.

Participants first watched an instructional video made by the Principal Investigator on how to pass a 9-0 nylon suture needle, and how to perform a microsurgical tie for a linear incision in a silicon baking mat using the same materials as would be provided to them for the pre- and post-assessments (Video 1). After watching the video three consecutive times, participants were tasked to pass and tie a 9-0 nylon suture in the same manner as the video recording. Their attempt at performing the microsurgical task was video-recorded for a pre-assessment with a cellphone camera focusing on the microscope field ensuring a clear view of the surgical field and the participant's instrument manipulation. Each subject wore gloves during the assessment to ensure anonymity.

After completion of the video-recorded pre-assessment, participants were randomized by flip of a coin to either the intervention group to build a micro-stellated icosahedron, or to the non-intervention control group with no assigned task. All subjects in both groups were required to return in two weeks for a second in-person meeting. At the second meeting, they were presented with the same instructional video as in the first meeting on how to pass a needle and perform a microsurgical tie. After watching the video three consecutive times, their attempt at completing a microsurgical tie was video-recorded for a post-assessment, using similar instruments and set-up as those used two weeks prior. Subjects in the intervention group were asked to return borrowed materials and their completed micro-stellated icosahedrons.

After all subjects were recruited, and their corresponding microsurgical tasks were video-recorded for pre- and post-assessments, each of the videos was edited to mute all audio in order to ensure anonymity. Each of the videos was de-identified by naming it with a random number from 1 to 42 and saved in a file folder in random order. This file folder was sent separately to two ophthalmologists, masked to the identity of the subjects (intervention vs control) and time of recording (pre- or post-assessment).

The raters used the Video-based Modified Objective Structure Assessment of Technical Skill (OSATS) Scoring Criteria, which scores four criteria with scores from 1 to 5: Economy of Movement, Confidence of Movement, Respect for Materials, and Precision of Operative Technique.4 The raters assigned separate scores for the participant's attempt at passing the needle through the incision, and for their attempt at tying a microsurgical tie. The attempt at passing the needle (Pass: Total) had a maximum possible score of 20, and the attempt at tying a microsurgical tie (Tie: Total) had a maximum possible score of 20, making 40 the maximum possible total score for each video (Total: Pass+Tie). The time each subject took to pass the needle, and the time each subject took to attempt tying a microsurgical tie was measured in number of seconds.

ELIGIBILITY:
Inclusion Criteria:

* 18 year-old or older.
* No prior microsurgical experience.

Exclusion Criteria:

* Prior microsurgical experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Change in Objective Structure Assessment of Technical Skill (OSATS) scores for passing a needle. | Two weeks
  The raters used the Video-based Modified Objective Structure Assessment of Technical Skill (OSATS) Scoring Criteria, which grades the following four criteria with a score from 1 (minimum) to 5 (maximum): Economy of Movement, Confidence of Movement, Respect for Materials, and Precision of Operative Technique. Therefore, by adding the grades for each of the four criteria, the total score for passing the needle (Pass: Total) had a minimum score of 4 and a maximum possible score of 20. Higher values represent better outcomes.
  Both raters assigned scores for the participants' attempts at passing the needle through the incision in each video. The scores from the two raters were added. The sum of the scores were used to determine whether there was change in scores for each participant between pre-assessment and post-assessment videos. Higher scores represent a better outcome.
Change in Objective Structure Assessment of Technical Skill (OSATS) scores for making a microsurgical tie. | Two weeks
  The raters used the Video-based Modified Objective Structure Assessment of Technical Skill (OSATS) Scoring Criteria, which grades the following four criteria with a score from 1 (minimum) to 5 (maximum): Economy of Movement, Confidence of Movement, Respect for Materials, and Precision of Operative Technique. Therefore, by adding the grades for each of the four criteria, the total score for making a microsurgical tie (Tie: Total) had a minimum score of 4 and a maximum possible score of 20. Higher values represent better outcomes.
  Both raters assigned scores for the participants' attempts at making a microsurgical tie in each video. The scores from the two raters were added. The sum of the scores were used to determine whether there was change in scores for each participant between pre-assessment and post-assessment videos. Higher scores represent a better outcome.
Change in time required to pass a needle. | Two weeks
  The time (in seconds) each subject took to pass the needle was measured from the time subject started manipulating the needle holder and toothed forceps to the time the subject began tying maneuvers.
  The time (in seconds) was used to determine whether there was change in the amount of time each subject required to pass the needle between pre-assessment and post-assessment videos. Lower values represent better outcomes.
Change in time required to complete microsurgical tie. | Two weeks
  The time (in seconds) each subject took to attempt tying a microsurgical tie was measured from the time the subject started manipulations for tying to the time the subject completed the microsurgical tie.
  The time(in seconds) was used to determine whether there was change in the amount of time each subject required to make a microsurgical tie between pre-assessment and post-assessment videos. Lower values represent better outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sangita P Patel, MD, PhD, Principal Investigator — State University of New York at Buffalo
Locations (1):
- Jacobs School of Medicine and Biomedical Sciences, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chan WY, Matteucci P, Southern SJ. Validation of microsurgical models in microsurgery training and competence: a review. Microsurgery. 2007;27(5):494-9. doi: 10.1002/micr.20393. PMID 17596849
- [Background] Dumestre D, Yeung JK, Temple-Oberle C. Evidence-based microsurgical skill-acquisition series part 1: validated microsurgical models--a systematic review. J Surg Educ. 2014 May-Jun;71(3):329-38. doi: 10.1016/j.jsurg.2013.09.008. Epub 2014 Jan 4. PMID 24797848
- [Background] Ericsson KA. Deliberate practice and the acquisition and maintenance of expert performance in medicine and related domains. Acad Med. 2004 Oct;79(10 Suppl):S70-81. doi: 10.1097/00001888-200410001-00022. No abstract available. PMID 15383395
- [Background] Ezra DG, Aggarwal R, Michaelides M, Okhravi N, Verma S, Benjamin L, Bloom P, Darzi A, Sullivan P. Skills acquisition and assessment after a microsurgical skills course for ophthalmology residents. Ophthalmology. 2009 Feb;116(2):257-62. doi: 10.1016/j.ophtha.2008.09.038. Epub 2008 Dec 16. PMID 19091411
- [Background] Benjamin L. Selection, teaching and training in ophthalmology. Clin Exp Ophthalmol. 2005 Oct;33(5):524-30. doi: 10.1111/j.1442-9071.2005.01089.x. PMID 16181283
- [Background] Belykh E, Byvaltsev V. Off-the-job microsurgical training on dry models: Siberian experience. World Neurosurg. 2014 Jul-Aug;82(1-2):20-4. doi: 10.1016/j.wneu.2014.01.018. Epub 2014 Feb 2. PMID 24495474
- [Background] White CA, Wrzosek JA, Chesnutt DA, Enyedi LB, Cabrera MT. A novel method for teaching key steps of strabismus surgery in the wet lab. J AAPOS. 2015 Oct;19(5):468-70.e1. doi: 10.1016/j.jaapos.2015.05.020. PMID 26486033
- [Background] Sikder S, Tuwairqi K, Al-Kahtani E, Myers WG, Banerjee P. Surgical simulators in cataract surgery training. Br J Ophthalmol. 2014 Feb;98(2):154-8. doi: 10.1136/bjophthalmol-2013-303700. Epub 2013 Oct 24. PMID 24158838
- [Background] Nandigam K, Soh J, Gensheimer WG, Ghazi A, Khalifa YM. Cost analysis of objective resident cataract surgery assessments. J Cataract Refract Surg. 2015 May;41(5):997-1003. doi: 10.1016/j.jcrs.2014.08.041. PMID 26049832
- [Background] McCannel CA. Continuous Curvilinear Capsulorhexis Training and Non-Rhexis Related Vitreous Loss: The Specificity of Virtual Reality Simulator Surgical Training (An American Ophthalmological Society Thesis). Trans Am Ophthalmol Soc. 2017 Aug 22;115:T2. eCollection 2017 Aug. PMID 29021716
- [Background] McCannel CA, Reed DC, Goldman DR. Ophthalmic surgery simulator training improves resident performance of capsulorhexis in the operating room. Ophthalmology. 2013 Dec;120(12):2456-2461. doi: 10.1016/j.ophtha.2013.05.003. Epub 2013 Jun 21. PMID 23796766
- [Background] Shrout PE, Fleiss JL. Intraclass correlations: uses in assessing rater reliability. Psychol Bull. 1979 Mar;86(2):420-8. doi: 10.1037//0033-2909.86.2.420. PMID 18839484
- [Background] Rufer F, Schroder A, Erb C. White-to-white corneal diameter: normal values in healthy humans obtained with the Orbscan II topography system. Cornea. 2005 Apr;24(3):259-61. doi: 10.1097/01.ico.0000148312.01805.53. PMID 15778595
- [Background] Lannon DA, Atkins JA, Butler PE. Non-vital, prosthetic, and virtual reality models of microsurgical training. Microsurgery. 2001;21(8):389-93. doi: 10.1002/micr.21709. PMID 11757067
- [Derived] Greyner-Almeida HD, Mahdavi Fard A, Chen C, Zhao J, Patel SP. A portable, low-cost practice model for microsurgical skills training. Int Ophthalmol. 2022 Aug;42(8):2323-2333. doi: 10.1007/s10792-022-02229-1. Epub 2022 Jan 29. PMID 35094230